CLINICAL TRIAL: NCT03622411
Title: The Effect of a Tablet-based Aphasia Therapy in the Chronic Phase After Stroke
Brief Title: Tablet-based Aphasia Therapy in the Chronic Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC/2018/0909
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Aphasia; Stroke
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aphasia therapy + speech app (Experimental): 3 hours per week of conventional aphasia therapy during 3 weeks + 5 hours per week during 3 weeks independent practice via the speech app
  Interventions: Device: speech app; Behavioral: aphasia therapy
- aphasia therapy + brain games (Active Comparator): 3 hours per week of conventional aphasia therapy during 3 weeks + 5 hours per week during 3 weeks of recreational tables use (brain games)
  Interventions: Device: brain games; Behavioral: aphasia therapy
- aphasia therapy (Active Comparator): 3 hours per week of conventional aphasia therapy during 3 weeks
  Interventions: Behavioral: aphasia therapy

INTERVENTIONS:
Device: speech app — language exercises provided by the speech therapist in hospital + independent practice of language exercises via a tablet and speech app
  Arms: aphasia therapy + speech app
Device: brain games — language exercises provided by the speech therapist in hospital + independent recreational tablet use via brain games
  Arms: aphasia therapy + brain games
Behavioral: aphasia therapy — language exercises provided by the speech therapist in hospital

SUMMARY:
Aphasia is one of the most common and disabling disorders following stroke, in many cases resolving in long-term deficits. There is evidence that intensive aphasia therapy is effective for language recovery, even in the chronic phase post-stroke. However, as many patients are left with residual language disorders and intensive aphasia rehabilitation is difficult to achieve, the investigators are exploring tablet-based therapies to further facilitate language recovery in a cost-effective manner.

DETAILED DESCRIPTION:
This study will investigate the clinical effects of intensive tablet-based aphasia therapy as an add-on to conventional aphasia therapy (= high intensive) compared to conventional aphasia therapy (either alone, or in combination with recreational tablet use (= low intensive) in patients with aphasia following stroke, as measured by specific linguistic tests, within task improvements, functional communication and quality of life.

Furthermore, the investigators want to learn more about the recovery of specific underlying language processes via event-related potentials (ERPs). At last, the investigators aim to explore whether patients with aphasia are satisfied with a tablet-based aphasia therapy, whether the app is user-friendly and which barriers the participants might have encountered.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with mild-severe aphasia (token test score between 7 and 49) after a left hemispheric ischemic or hemorrhagic stroke
* inclusion starting from 6 months post-stroke
* age 18 - 85 years
* being right-handed (according to the questionnaire for handedness, Van Strien)
* mother tongue: Dutch
* imaging (CT or MRI) prior to inclusion
* signed informed consent

Exclusion Criteria:

* history of a previous stroke with persistent (> 24 hours) language symptoms
* history of other diseases of the central nervous system, psychological disorders and (developmental) speech and/or language disorders
* serious non-linguistic, cognitive disorders (as documented in the patients' medical history)
* inability to perform tablet-based tasks (based on a short training session)
* excessive use of alcohol or drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Boston Naming Test (BNT) | 4 months
  Measure of word retrieval. Patients will have to name line drawings that gradually increase in difficulty

SECONDARY OUTCOMES:
Spontaneous speech of the Aachen Aphasia Test (AAT) | 4 months
  spontaneous speech is elicited and scored during a semi-standardized interview
Quality of life (SAQOL-39-Nl) | 4 months
  a questionnaire investigating the health-related quality of life of patients following stroke
Usability questionnaire | 1 day
  a self-prepared 5 point-Likert Scale concerning the usability of the app

CONTACTS AND LOCATIONS:
Overall Officials: Veerle De Herdt, Principal Investigator — University Ghent
Locations (1):
- University Hospital, department of neurology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided